CLINICAL TRIAL: NCT00608751
Title: A Feasibility Study of Adaptive Intensity-Modulated Radiation Therapy in the Definitive Treatment of Head-and-Neck Cancer
Brief Title: A Feasibility Study of Adaptive Intensity-Modulated Radiation Therapy
Acronym: IMRT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of accrual and software issues
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1210
Record Dates: First submitted 2008-01-02; First posted 2008-02-06 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Head and Neck Cancer
Keywords: Newly Diagnosed head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT (Experimental): External beam radiation with 6 MV photons will be delivered in 200 cGy daily fractions, 35 fractions over 7 weeks for a total dose of 7000 cGy.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT

SUMMARY:
Patients with head and neck cancer and are schedule to receive standard radiation therapy known as IMRT to treat cancer

DETAILED DESCRIPTION:
In this study, we will plan additional measurements of the position of the patient's organs weekly during radiation treatment. We will analyze these measurements in order to evaluate whether we need to adjust our treatment procedures for the remainder of the treatments. We might adjust the dose of radiation received to specific organs in order to try to minimize the amount of radiation the healthy tissue receives.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Karnofsky Performance Status of >= 60
* New diagnosis of head-and-neck cancer, all subsites included (i.e. nasopharynx, oropharynx, oral cavity, hypopharynx, larynx.)
* All stages with measurable gross disease (>= 1.0 cm) by CT imaging
* Pathologic confirmation of squamous cell carcinoma by biopsy or cytology
* Signed study-specific consent form
* Sequential or concurrent chemotherapy is allowed but not mandated. (no chemotherapy is allowed if patient is judged not to be a candidate for chemotherapy by the medical oncologist)

Exclusion Criteria

* Age < 18
* Karnofsky Performance Status < 60
* Radiographic or pathologic evidence of distant metastatic disease (i.e. other than cervical lymph nodes)
* Prior radiation therapy to the head-and-neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of adaptive radiation therapy in the definitive treatment (MLC-based IMRT or helical tomotherapy) | 7 weeks
  Feasibility is determined by employing weekly 3D onboard imaging for plan re-evaluation and initiation of an adaptive process if the original PTV and/or normal structure goals are compromised.

SECONDARY OUTCOMES:
Measure additional time required by physician and ancillary staff for the process of adaptive IMRT | 7 weeks
  Recording on a weekly basis the actual time required for repeat CT imaging, plan re-evaluation, replanning, and repeat physics QA.
Identify a subset of patients in whom adaptive IMRT would be recommended | 7 weeks
Measure acute and late toxicity | Until patient death
Local, regional, and distant recurrence | Until recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Wade Thorstad, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu